CLINICAL TRIAL: NCT04198584
Title: Pilot Feasibility Testing of a Small Randomized Controlled Trial to Evaluate a Telemedicine Stress Management and Lifestyle Group Intervention for Patients With Symptomatic Chronic Hepatitis C
Brief Title: Study of Telemedicine Stress Management and Lifestyle Group Intervention for HCV Patients
Acronym: VC-CBCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-2197; 1R21NR017908-01A1 (NIH)
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2021-05

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: Participants (n=32) were assigned by 3:1 randomization to VC-CBCS or SC. Participants were recruited in 4 cohorts (Wave 1: n=7, Wave 2: n=9, Waves 3, 4: n=8 each). In Wave 1, 5 participants were randomized to VC-CBCS and 2 to SC. In Wave 2, 7 participants were randomized to VC-CBCS and 2 to SC. In Waves 3 and 4, 6 participants were randomized to VC-CBCS and 2 to SC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VC-CBCS Intervention (Experimental): The VC-CBCS intervention was delivered via WebEx videoconferencing technology and included 14, 2-hour long sessions that involved group-based psychoeducation, cognitive and behavioral skills training, stress management, relaxation practice and healthy lifestyle habits to support overall health and liver health. Intervention materials included a hard copy Patient Workbook and audio-recorded relaxation techniques.
  Interventions: Behavioral: VC-CBCS
- Standard of Care (SC) (No Intervention): Participants randomized to SC received no intervention and were followed by medical providers in clinic per clinical practice guidelines and clinicians discretion.

INTERVENTIONS:
Behavioral: VC-CBCS — A 14-module stress management and lifestyle group-based intervention delivered via videoconferencing WebEx technology to participants who have/had chronic hepatitis C and experience symptoms, stress or lifestyle requirements to promote liver health.
  Arms: VC-CBCS Intervention

SUMMARY:
A pilot feasibility study of a small randomized controlled trial (RCT) comparing a video-conferencing cognitive behavioral coping skills (VC-CBCS) group to standard of care (SC) for symptomatic patients previously diagnosed with chronic hepatitis C to evaluate feasibility, patient satisfaction and differences in symptoms, quality of life and liver markers.

DETAILED DESCRIPTION:
This is a pilot feasibility study of a small randomized controlled trial (RCT) to evaluate a cognitive behavioral coping skills (CBCS) delivered via videoconferencing, referred to as the "VC-CBCS" compared to standard of care (SC). The study included a representative sample of 32 symptomatic patients who have/had chronic hepatitis C. Patients (n=32) were randomized in a 1:3 ratio to (1) standard of care (SC) or (2) to participate in 14, two hour VC-CBCS sessions. Four groups of patients were randomized and consisted of 7-9 patients each. The groups were as follows:

* Group 1: 7 patients with 5 randomized to VC-CBCS and 2 to SC;
* Group 2: 9 patients with 7 randomized to VC-CBCS and 2 to SC;
* Groups 3 and 4: 8 patients each with 6 randomized to VC-CBCS and 2 to SC each group.

Each wave of VC-CBCS patients formed a group to join the Group Facilitator via a WebEx platform on a weekly basis using iPads from their homes. The telehealth intervention provided group-based education, skills and practices involving stress management, coping with symptoms, and support for healthy lifestyle changes. The researchers examined: (1) the feasibility of delivering a group intervention via telehealth technology remotely using iPads, (2) participant satisfaction with the intervention, and (3) whether differences are observed in several outcomes between the two conditions on quality of life, physical and mental symptoms, and liver markers. Participants completed patient-reported outcome (PRO) surveys at four time points during the study, with main outcomes being change from pre-intervention to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older;
* Medically cleared by hepatology
* Patients who are currently or were previously diagnosed with chronic Hepatitis C Viral (HCV) infection;
* Evidence of ongoing symptoms, stress, or unhealthy lifestyle habits, defined as a score of greater than or equal to 4 on a scale 0(none) - 10 (severe) on two or more numeric rating scale questions (see Screening Form 1);
* Able to read and speak English.

Exclusion Criteria:

* Decompensated liver disease (Childs Pugh C) judged by hepatologist or recorded in patient medical record;
* Life expectancy of <12 months estimated by hepatologist;
* Has had a liver transplant or is on the wait list for a transplant
* Severe alcohol or substance use disorder, psychiatric disorder or cognitive impairment that is likely to interfere with the ability to participate in telehealth groups and follow guidelines about group participation as judged by the Hepatology provider or research staff;
* Lack of private, quiet space in home in which to participate in VC-CBCS sessions
* Unwilling to have intervention sessions audio-recorded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna M. Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 participants were approached for study interest; 39 were consented and of those 32 were enrolled.
Groups:
- VC-CBCS Intervention: The VC-CBCS intervention was delivered via WebEx videoconferencing technology and included 14, 2-hour long sessions that include group-based psychoeducation, cognitive and behavioral skills training, stress management, relaxation practice and healthy lifestyle habits to support overall health and liver health. Intervention materials included a hard copy Patient Workbook and audio-recorded relaxation techniques.
- Standard of Care (SC): Participants randomized to Standard of Care (SC) received no intervention and were followed by medical providers in clinic per clinical practice guidelines and clinicians discretion.
Period: Overall Study
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Started | 24 | 8
Randomized to Wave 1 | 5 | 2
Randomized to Wave 2 | 7 | 2
Randomized to Wave 3 | 6 | 2
Randomized to Wave 4 | 6 | 2
Total Randomized | 24 | 8
Actually Received Treatment | 21 | 8
Completed | 19 | 8
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- VC-CBCS Intervention: The VC-CBCS intervention was delivered via WebEx videoconferencing technology and included 14, 2-hour long sessions that included group-based psychoeducation, cognitive and behavioral skills training, stress management, relaxation practice and healthy lifestyle habits to support overall health and liver health. Intervention materials included a hard copy patient Workbook and audio-recorded relaxation techniques.
- Total: Total of all reporting groups
Arm/Group | VC-CBCS Intervention | Standard of Care (SC) | Total
Number analyzed (Participants) | 24 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7.5) | 56 (11.4) | 56 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 19 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was patient-reported on the T1 baseline surveys by patients who were enrolled and completed their T1 surveys.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 14 | 5 | 19
    Unknown or Not Reported | 10 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 16 | 5 | 21
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Consented Versus Approached
Description: One feasibility measure was to evaluate the percentage of patients consented compared to those approached for participation in the study.
Time Frame: Six Months
Measure: Number; unit: percentage of participants
Groups:
- All Patients: All patients who were approached for the study.
Arm/Group | All Patients
Number analyzed (Participants) | 53
percentage of participants | 74

2. Primary Outcome: Percentage of Participants Consented Versus Randomized
Description: One feasibility measure was to evaluate the percentage of participants randomized for the study compared to those consented.
Time Frame: Six Months
Measure: Number; unit: percentage of participants
Groups:
- All Participants: All participants who were consented for the study.
Arm/Group | All Participants
Number analyzed (Participants) | 39
percentage of participants | 82

3. Primary Outcome: Percentage of Standard of Care Condition Participants Retained vs Enrolled
Description: Percentage of standard of care condition participants retained in the study compared to those enrolled. Retention is defined as participants who submitted PRO assessments up through T4 (end of study).
Time Frame: Six Months
Measure: Number; unit: percentage of participants
Groups:
- Standard of Care (SC): Participants randomized to SC received no intervention and were followed by medical providers in clinic per clinical practice guidelines and clinicians' discretion. Participants completed survey assessments four times during the study.
Arm/Group | Standard of Care (SC)
Number analyzed (Participants) | 8
percentage of participants | 100

4. Primary Outcome: Percentage of VC-CBCS Intervention Condition Participants Retained vs Enrolled
Description: Percentage of VC-CBCS Intervention participants retained in the study compared to those enrolled. Retention is defined as participants who completed at least 3 intervention sessions.
Time Frame: Six Months
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention
Number analyzed (Participants) | 24
percentage of participants | 79.2

5. Primary Outcome: Percentage of Surveys Completed by Participants Who Completed the Study
Description: Percentage of surveys over time completed by participants who completed the study. Surveys included 12 patient-reported primary and secondary outcome measures. Completion was defined as submission of each of the 12 surveys at Time 1 (T1) through Time 4 (T4).
Time Frame: Baseline (T1) to Week 14 (T4)
Population: Data collection rate is for those who completed the study - 8 Standard of Care and 19 VC-CBCS, total of 27 participants.
Measure: Number; unit: percentage of surveys completed
Groups:
- All Enrolled Participants: All participants who were enrolled and completed the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 27
percentage of surveys completed | 99.4

6. Primary Outcome: Global Health Status Physical Health Mean T-Score
Description: The Patient Reported Outcome Measurement Information System (PROMIS) Global Health Status measure is a 10-item short form that was used to measure an individual's physical, mental, and social health. Item responses range from 5 = None to 1 = Very Severe. The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 16.2 to 67.7. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation better (more healthy) than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 45.7 [27.3 to 64.1] | 41.8 [27.2 to 56.4]
  Week 14 (T4) | 46.0 [31.7 to 60.3] | 48 [31.5 to 64.5]

7. Primary Outcome: Global Health Status Mental Health Mean T-Score
Description: The PROMIS Global Health Status measure is a 10-item short form that was used to measure an individual's physical, mental, and social health. Item responses range from 5 = None to 1 = Very Severe. The adult PROMIS Global Health measure produces two scores: Physical Health and Mental Health. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 21.2 to 67.7. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation better (more healthy) than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 46.7 [27.7 to 65.7] | 41.9 [26.0 to 57.8]
  Week 14 (T4) | 49.3 [34.6 to 64.0] | 45.9 [31.0 to 60.8]

8. Primary Outcome: Depression Mean T-score
Description: The PROMIS Depression measure is an 8-item short form that was used to measure patient-reported depression. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 41.0 to 79.4. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more (more Depression) than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- VC-CBCS Intervention: The VC-CBCS intervention was delivered via WebEx videoconferencing technology and included 14, 2-hour long sessions that included group-based psychoeducation, cognitive and behavioral skills training, stress management, relaxation practice and healthy lifestyle habits to support overall health and liver health. Intervention materials included a hard copy Patient Workbook and audio-recorded relaxation techniques.
  VC-CBCS: A 14 module stress management and lifestyle group-based intervention delivered via videoconferencing Webex technology to patients who have had chronic hepatitis C and experience symptoms, stress or lifestyle requirements to promote liver health.
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 52.3 [35.2 to 69.4] | 51.6 [31.0 to 72.2]
  Week 14 (T4) | 48.6 [35.1 to 62.1] | 49.0 [33.0 to 65.0]

9. Primary Outcome: Anger Mean T-score
Description: The PROMIS Anger measure is a 5-item short form that was used to measure patient-reported anger. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 32.9 to 82.9. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more Anger and T-score=40 is 1 standard deviation less Anger than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 51.0 [31.8 to 70.2] | 52.3 [31.3 to 73.3]
  Week 14 (T4) | 46.5 [30.8 to 62.2] | 46.9 [26.8 to 67.0]

10. Primary Outcome: Anxiety Mean T-score
Description: The PROMIS Anxiety measure is a 4-item short form that was used to measure patient-reported anxiety. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 40.3 to 81.6. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more Anxiety and T-score=40 is 1 standard deviation less Anxiety than the general population. The Anxiety T-score can range from 40.3 - 81.6.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 52.7 [33.9 to 71.5] | 57.7 [42.0 to 73.4]
  Week 14 (T4) | 50.4 [34.7 to 66.1] | 51.2 [34.6 to 67.8]

11. Primary Outcome: Fatigue Mean T-score
Description: The PROMIS Fatigue measure is a 7-item short form that was used to measure patient-reported fatigue. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 29.4 to 83.2. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more Fatigue and T-score=40 is 1 standard deviation less Fatigue than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 51.9 [30.4 to 73.4] | 50.4 [30.5 to 70.3]
  Week 14 (T4) | 48.6 [29.9 to 67.3] | 46.6 [26.6 to 66.6]

12. Primary Outcome: Sleep Disturbance Mean T-score
Description: The PROMIS Sleep Disturbance measure is an 8-item short form that was used to measure patient-reported sleep disturbance. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 32.0 to 73.3. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more Sleep Disturbance and T-score=40 is 1 standard deviation less Sleep Disturbance than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 52.0 [33.4 to 70.6] | 50.8 [37.6 to 64.0]
  Week 14 (T4) | 50.0 [36.6 to 63.4] | 46.0 [26.6 to 65.4]

13. Primary Outcome: Pain Interference Mean T-score
Description: The PROMIS Pain Interference measure is an 8-item short form that was used to measure patient-reported pain interference. Item responses range from 1 = Never to 5 = Always. The raw scores are converted into a T-score. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. The minimum and maximum T-scores ranged from 41.6 to 75.6. Higher T- scores indicate more of that construct, for example, a T-score=60 is 1 standard deviation more Pain Interference and T-score=40 is 1 standard deviation less Pain Interference than the general population.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
T-score
  Baseline (T1) | 53.5 [37.0 to 70.0] | 55.8 [39.9 to 71.7]
  Week 14 (T4) | 52.0 [34.6 to 69.4] | 54.6 [37.5 to 71.7]

14. Secondary Outcome: Perceived Stress Mean Score
Description: The Perceived Stress Scale (PSS) is a widely used survey to measure stress perception. The scale includes 10 items, rated using a 5-point scale, from 0 (never) to 4 (very often) where patients report the frequency of stress symptoms in the past month. Items are summed with a minimum and maximum ranging from 0 to 40. Higher PSS scores reflect higher subjective stress.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 24.2 [20.8 to 27.7] | 23.9 [18.9 to 28.9]
  Week 14 (T4) | 20.6 [17.9 to 23.4] | 21.8 [16.1 to 27.4]

15. Secondary Outcome: Coping Skills Confidence Mean Score
Description: The Measure of Current Status (MOCS)-Part A measured participant confidence in performing multiple skills including stress awareness, relaxation, assertiveness, and coping skills. The scale contains 13 items rated on a scale from 0 = I cannot do this at all to 4 = I can do this extremely well. A Total Coping Skills score is created by taking the average of the 13 items. The Total Coping Skill score can range from a minimum of 0 to a maximum of 4.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 2.18 [1.8 to 2.6] | 2.16 [1.7 to 2.6]
  Week 14 (T4) | 2.74 [2.4 to 3.1] | 2.38 [1.9 to 2.9]

16. Secondary Outcome: Participant Satisfaction With VC-CBCS Intervention Mean Score
Description: After each VC-CBCS intervention session, participants completed a 14-item acceptability/satisfaction survey about their impressions with the current intervention session. Items are scored on a scale from 1= not at all to 5=extremely useful. Data across all VC-CBCS participants and all intervention sessions were averaged into a Total Patient Satisfaction score that could range from a minimum of 1 to a maximum of 5 with higher scores indicating greater satisfaction.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: Participants randomized to Standard of Care received no intervention and did not complete survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention
Number analyzed (Participants) | 19
score on a scale | 4.23 (0.5)

17. Secondary Outcome: Aspartate Aminotransferase (AST) Mean Score for Females
Description: Liver enzyme level (AST U/L). Reference range for females is 14-38 U/L. Numbers higher than these reference ranges are considered in the abnormal range and can suggest liver damage or inflammation. These comparisons were only made for participants who had already achieved viral cure at baseline and who were not on medical treatment for chronic hepatitis C at baseline.
Time Frame: Baseline (T1), Week 14 (T4)
Population: The analytic sample includes 4 females who completed the VC-CBCS intervention and 3 females in Standard of Care. Of these, 1 VC-CBCS Intervention participant had missing data at T4. Of the 3 females in Standard of Care, 2 had missing data at T1 and all 3 participants had missing data at T4.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 4 | 1
U/L
  Baseline (T1) | 28.0 (8.91) | 23.0 (0.0)
  Week 14 (T4): number analyzed (Participants) | 3 | 0
  Week 14 (T4) | 31.0 (8.89) |

18. Secondary Outcome: Aspartate Aminotransferase (AST) Mean Score for Males
Description: Liver enzyme level (AST U/L). Reference range for males is 19-55 U/L. Numbers higher than these reference ranges are considered in the abnormal range and can suggest liver damage or inflammation. These comparisons were only made for participants who had already achieved viral cure at baseline and who were not on Hepatitis C Virus (HCV) treatment at baseline.
Time Frame: Baseline (T1), Week 14 (T4)
Population: The analytic sample includes 14 males who completed the VC-CBCS intervention and 5 males in Standard of Care. Of these, 4 VC-CBCS Intervention participants had missing data at T1 and 5 at T4. Of the 5 males in Standard of Care, 1 had missing data at T1 and 2 had missing data at T4.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 11 | 4
U/L
  Baseline (T1) | 34.7 (11.2) | 36.5 (17.3)
  Week 14 (T4): number analyzed (Participants) | 10 | 3
  Week 14 (T4) | 30.0 (8.39) | 45.3 (31.8)

19. Secondary Outcome: Alanine Aminotransferase (ALT) Mean Score for Females
Description: Liver enzyme level (ALT U/L). Reference range for females is <35 U/L. Numbers higher than these reference ranges are considered in the abnormal range and can suggest liver damage or inflammation. These comparisons were only made for participants who had already achieved viral cure at baseline and who were not on HCV treatment at baseline.
Time Frame: Baseline (T1), Week 14 (T4)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 4 | 1
U/L
  Baseline (T1) | 22.0 (13.0) | 13.0 (0.0)
  Week 14 (T4): number analyzed (Participants) | 3 | 0
  Week 14 (T4) | 28.3 (20.0) |

20. Secondary Outcome: Alanine Aminotransferase (ALT) Mean Score for Males
Description: Liver enzyme level (ALT U/L). Reference range for males is <50 U/L. Numbers higher than these reference ranges are considered in the abnormal range and can suggest liver damage or inflammation. These comparisons were only made for participants who had already achieved viral cure at baseline and who were not on HCV treatment at baseline.
Time Frame: Baseline (T1), Week 14 (T4)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 11 | 4
U/L
  Baseline (T1) | 34.6 (23.0) | 33.0 (10.3)
  Week 14 (T4): number analyzed (Participants) | 10 | 3
  Week 14 (T4) | 36.9 (24.1) | 28.0 (12.5)

21. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Sleep Quality Mean Score
Description: Item 9 from the Pittsburgh Sleep Quality Index (PSQI) was used to measure sleep quality. All participants completed this measure at PRO time points T1 and T4 that covered 30 days prior to assessment. "During the past month, how would you rate your sleep quality overall?" The response set ranged from a minimum of 0 (Very Good) to a maximum of 3 (Very Bad). Higher scores indicated worse sleep quality.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 1 Standard of Care participant missing data for this variable at T4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 1.32 (0.82) | 1.13 (0.64)
  Week 14 (T4): number analyzed (Participants) | 19 | 7
  Week 14 (T4) | 1.05 (0.52) | 0.71 (0.76)

22. Secondary Outcome: Percentage of Overall Medication Adherence
Description: Medication Adherence Visual Analog Scales (VAS) was used to evaluate medication adherence for up to five daily medications for multiple comorbidities in the past 7 days in participants who were prescribed medications at baseline. Participants reported the average adherence over the course of 7 days for each medication on a scale from 0% to 100% adherence for each medication. The average percent adherence was created for all medications for each patient and could range from 0% to 100%. Overall medication adherence adherence was assessed at T1 and T4.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 7 VC-CBCS Intervention participants were excluded from the analysis because they were not prescribed daily medications at Baseline (T1). Two of the 12 VC-CBCS participants and 4 of the Standard of Care participants were missing data for this variable at T4.
Measure: Number (95% Confidence Interval); unit: percentage of medication adherence
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 12 | 8
percentage of medication adherence
  Baseline (T1) | 85.2 [73.9 to 96.5] | 96.9 [94.7 to 99.1]
  Week 14 (T4): number analyzed (Participants) | 10 | 4
  Week 14 (T4) | 92.8 [85.4 to 100.3] | 89.8 [72.6 to 106.9]

23. Secondary Outcome: Alcohol Total Mean Score
Description: Three items from the Substance Abuse and Mental Illness Symptoms Screener (SAMISS) Survey was administered at baseline (T1) and Week 14 (T4) to evaluate self-reported alcohol use in all participants. The three items evaluated frequency, amount of alcohol consumption, and binge drinking. Individual scores could range from 0 to 4, with higher scores indicating higher consumption.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 1 VC-CBCS Intervention participant with missing data at T1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1): number analyzed (Participants) | 18 | 8
  Baseline (T1) | 1.39 (2.43) | 0.13 (0.35)
  Week 14 (T4) | 0.95 (2.27) | 0.25 (0.71)

24. Secondary Outcome: Percentage of Participants Who Improved Fruit Consumption by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items assessed fruit intake as a health behavior - "Over the past 12 months, how often did you eat fruits?" Original 8-point response scale ranged from "1 time per month" to "2 or more times/day." Recoded 8 categories into 4 categories, ranging from "Daily consumption" to "Less than weekly". The percentage shown is the number of participants who improved by 1 or more categories based on the 4 category levels from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 1 Standard of Care participant missing data for this variable
Measure: Number; unit: percentage of patients
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 7
percentage of patients | 47.0 | 43.0

25. Secondary Outcome: Percentage of Participants Who Improved Vegetable Consumption by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured vegetable intake as a health behavior - "Over the past 12 months, how often did you eat vegetables?" Original 8-point response scale ranged from "1 time per month" to "2 or more times/day." Recoded 8 categories into 4 categories, ranging from "Daily consumption" to "Less than weekly". The percentage is the number of participants who improved by 1 or more categories on the 4 category levels from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 1 Standard of Care participant missing data for this variable
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 7
percentage of participants | 16 | 14

26. Secondary Outcome: Percentage of Participants Who Complete Moderate Activity for at Least 10 Minutes at a Time
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured moderate activity as a health behavior in all participants at T1 (baseline) and T4 (week 14) and will cover 30 days prior to assessment. BRFSS item asks "Do you do moderate activity for at least 10 minutes at a time"? Response options: Yes/No. Percentage is participants who indicate "Yes" to doing moderate activity for at least 10 minutes at a time
Time Frame: Baseline (T1), Week 14 (T4)
Population: 1 VC-CBCS Intervention participant with missing data at T1.
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
percentage of participants
  Baseline (T1): number analyzed (Participants) | 18 | 8
  Baseline (T1) | 73.7 | 50.0
  Week 14 (T4) | 78.9 | 87.5

27. Secondary Outcome: Mean Number of Minutes of Moderate Activity Per Week
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured moderate activity as a health behavior by combining two BRFSS items: "If yes, how many days per week do you do these moderate activities for at least 10 minutes at a time" and "If yes, how much total time per day do you spend doing these activities?" Total number of minutes of moderate activity per week calculated as number of days x number of minutes.
Time Frame: Baseline (T1) , Week 14 (T4)
Population: 5 participants with missing data for this variable (4 VC-CBCS intervention participants, 1 Standard of Care)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 15 | 7
minutes
  Baseline (T1) | 314 (556) | 87.9 (120)
  Week 14 (T4) | 528 (808) | 170 (257)

28. Secondary Outcome: Percentage of Participants Who Complete Vigorous Activity for at Least 10 Minutes at a Time
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured vigorous activity as a health behavior - BRFSS Item "Do you do vigorous activity for at least 10 minutes at a time?" Response option: Yes/No. Percentage is participants who indicate "Yes" to doing vigorous activity for at least 10 minutes at a time
Time Frame: Baseline (T1), Week 14 (T4)
Population: 1 VC-CBCS Intervention participant missing data for this variable
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 18 | 8
percentage of participants
  Baseline (T1) | 42.1 | 50.0
  Week 14 (T4) | 47.4 | 25.0

29. Secondary Outcome: Mean Number of Minutes of Vigorous Activity Per Week
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured vigorous activity as a health behavior by combining two BRFSS items: "If yes, How many days per week do you do these vigorous activities for at least 10 minutes at a time" and "If yes, how much total time per day do you spend doing these activities?" Total number of minutes of vigorous activity per week calculated as number of days x number of minutes.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 2 participants missing data for this variable (1 VC-CBCS Intervention, 1 Standard of Care)
Measure: Mean (Standard Deviation); unit: total minutes in a week
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 18 | 7
total minutes in a week
  Baseline (T1) | 241 (457) | 55.7 (74.4)
  Week 14 (T4) | 235 (513) | 17.1 (34.0)

30. Secondary Outcome: Mean Time Spent Sitting on the Weekdays
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured sedentarism as a health behavior - BRFSS item "What is the total number of hours you spend siting on a weekday?" The mean can range from a minimum of 0 to maximum of 24 hours. Average numbers of hours spent sitting on the weekday was assessed at T1 to T4.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 1 Standard of Care participant missing data for this variable
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 7
hours
  Baseline (T1) | 8.95 (3.44) | 6.57 (4.08)
  Week 14 (T4) | 7.0 (2.28) | 7.0 (2.31)

31. Secondary Outcome: Mean Time Spent Sitting on the Weekends
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured sedentarism as a health behavior - BRFSS Item "What is the total number of hours you spend sitting on a weekend day?" Mean ranges from a minimum of 0 to maximum of 24 hours. Average numbers of hours spent sitting on the weekends assessed at T1 and T4.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
hours
  Baseline (T1) | 7.68 (3.53) | 6.0 (3.66)
  Week 14 (T4) | 4.22 (2.26) | 6.43 (3.10)

32. Secondary Outcome: Percentage of Participants Who Reduced Regular Soda Intake by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured soda intake as a health behavior - BRFSS item "During the past 30 days, how often did you drink regular soda or pop that contains sugar? Do not include diet soda or diet pop." Original 9-point response scale ranged from "Never" to "6 more more per day." Recoded 9 categories into 5 categories, ranging from "Never" to Daily." The percentage is the number of participants who improved (consumed less) by 1 or more categories on the 5 category levels from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 3 participants missing data for this variable (2 VC-CBCS Intervention participants, 1 Standard of Care participant)
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 17 | 7
percentage of participants | 35 | 14

33. Secondary Outcome: Percentage of Participants Who Reduced Diet Soda Intake by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured diet soda intake as a health behavior - BRFSS item "During the past 30 days, how often did you drink diet soda or diet pop that contains an artificial sweeter?" Original 9-point response scale ranged from "Never" to "6 or more per day." Recoded 9 categories into 5, ranging from "Never" to Daily." The percentage is the number of patients who improved (consumed less) by 1 or more categories on the 5 recoded category level from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 2 Standard of Care participants missing data for this variable
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 6
percentage of participants | 5 | 17

34. Secondary Outcome: Percentage of Participants Who Reduced Fruit Juice Intake by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured fruit juice intake as a health behavior - BRFSS item "During the past month, how many times per day, week or month did you drink 100% pure fruit juices? Original 9-point response scale ranged from "Never" to "6 or more per day." Recoded 9 categories into 5, ranging from "Never" to Daily." The percentage is the number of participants who improved (consumed less) by 1 or more categories on the 5 recoded category levels from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 1 Standard of Care participant missing data for this variable
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 7
percentage of participants | 16 | 29

35. Secondary Outcome: Percentage of Participants Who Reduced Meals From Fast Food Restaurants by One or More Categories
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured fast food intake as a health behavior - BRFSS item "In a typical week, how many of your own meals come from fast food restaurants?" Original 9-point response scale ranged from "Never" to "6 or more per day." Recoded 9 categories into 5, ranging from "Never" to Daily." The percentage is the number of participants who improved (reduced) by 1 or more categories on the 5 recoded category levels from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 3 participants were missing data for this variable (1 VC-CBCS Intervention participant, 2 Standard of Care participants)
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 18 | 6
percentage of participants | 39 | 17

36. Secondary Outcome: Percentage of Participants Who Increased Dinners Prepared at Home by 1 or More Days
Description: Behavioral Risk Factor Surveillance System (BRFSS) items measured food prepared at home as a health behavior - BRFSS item "On how many days per week do you usually eat a dinner that is prepared at home?" 7-point response scale ranged from 0 to 7 days. The percentage is the number of patients who improved (increased) by 1 or more days from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: Three participants were missing data for this variable (2 VC-CBCS Intervention participants, 1 Standard of Care participant)
Measure: Number; unit: percentage of participants
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 17 | 7
percentage of participants | 35 | 0

37. Secondary Outcome: Change in Weight (Lbs)
Description: Change in weight (lbs) among those who had pre-intervention BMI > 24.9 (obese and above) from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 8 participants had missing data for this variable (4 VC-CBCS Intervention, 4 Standard of Care)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 15 | 4
pounds | -2.67 (13.7) | 0.0 (3.56)

38. Secondary Outcome: Change in Percent Weight Change
Description: Change in percent weight (lbs) among those who had pre-intervention BMI > 24.9 (obese and above) from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 8 participants had missing data for this variable (4 VC-CBCS Intervention, 4 Standard of Care)
Measure: Mean (Standard Deviation); unit: percent of weight change
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 15 | 4
percent of weight change | 0.91 (5.65) | -0.23 (1.91)

39. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in Body Mass Index (BMI) among those who had pre-intervention BMI > 24.9 (obese and above) from T1 to T4.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: 8 participants had missing data for this variable (4 VC-CBCS Intervention, 4 Standard of Care)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 15 | 4
kg/m^2 | -0.53 (2.28) | 0.23 (0.83)

40. Secondary Outcome: Prescription Drug Misuse Total Mean Score
Description: Surveys administered at baseline (T1) and Week 14 (T4) evaluated self-reported prescription drug misuse in all participants. One item from the Substance Abuse and Mental Illness Symptoms Screener (SAMISS) Survey evaluated misuse of prescription drugs in the last year. The response options ranged from a minimum of 0="Never" to a maximum of 4="Daily/Almost Daily". Higher scores indicate higher consumption.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 0.11 (0.32) | 0.0 (0.0)
  Week 14 (T4) | 0.11 (0.32) | 0.0 (0.0)

41. Secondary Outcome: Non-prescription Street Drug Use Total Mean Score
Description: Surveys administered at baseline (T1) and Week 14 (T4) evaluated self-reported non-prescription street drug use in all participants. One item from the Substance Abuse and Mental Illness Symptoms Screener (SAMISS) Survey evaluated non-prescription street drug use in the last year. The response options ranged from a minimum of 0="Never" to a maximum of 4="Daily/Almost Daily". Higher scores indicate higher consumption.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 1.37 (1.71) | 0.88 (1.36)
  Week 14 (T4) | 0.95 (1.47) | 0.13 (0.35)

42. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Sleep Efficiency Composite Mean Score
Description: Items 1, 3 and 4 from the Pittsburgh Sleep Quality Index (PSQI) were used to create a Sleep Efficiency composite score. All participants completed this measure at T1 and T4 that covered 30 days prior to assessment. The sleep efficiency score = (# hours slept/# hours in bed) X 100% .The sleep efficiency composite score ranged from: 0 = >85% efficiency,
  1 = 75-84% efficiency, 2= 65-74% efficiency, and 3= <65%. Lower scores indicate better sleep efficiency.
Time Frame: Baseline (T1), Week 14 (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 1.05 (1.22) | 1.38 (1.30)
  Week 14 (T4) | 1.26 (1.37) | 0.75 (1.04)

43. Secondary Outcome: Healthy Sleep Behaviors Mean Score
Description: One item "In the last month, how often did you engage in healthy sleep behaviors before bedtime?" evaluated healthy sleep behaviors. All participants completed this measure at T1 and T4. The response set ranged from 0 (not at all) to 4 (almost every night). Higher scores indicated better sleep behaviors.
Time Frame: Baseline (T1), Week 14 (T4)
Population: 2 Standard of Care participants were missing data for this variable at T4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 19 | 8
score on a scale
  Baseline (T1) | 1.37 (1.26) | 2.13 (0.99)
  Week 14 (T4): number analyzed (Participants) | 19 | 6
  Week 14 (T4) | 2.42 (0.84) | 2.17 (1.33)

44. Other Pre Specified Outcome: Salivary Cortisol Area Under the Curve With Respect to Ground (AUC-G)
Description: Participants in both conditions collected saliva samples at Baseline (T1) and Week 14 (T4). Participants were instructed to collect four saliva samples at each timepoint; 1) immediately upon awakening 2) 30 minutes after awakening 3) late afternoon 4) before bedtime. The mean AUC-G was then obtained at T1 and T4. Mean AUC-G scores could range from 0.195 to 2.29.
Time Frame: Baseline (T1), Week 14 (T4)
Population: T1: Data from 1 Standard of Care participant were excluded due to nontraditional sleep schedule. Data from 5 VC-CBCS Intervention participants were excluded due to missing data, nontraditional sleep schedules, and/or noncompliance with sample collection instructions.
  T4: Data from 2 Standard of Care participants and 7 VC-CBCS Intervention participants were excluded due to missing data, nontraditional sleep schedules, and/or noncompliance with sample collection instructions.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
Number analyzed (Participants) | 14 | 7
ug/dL
  Baseline (T1) | 1.01 (0.54) | 1.18 (0.65)
  Week 14 (T4): number analyzed (Participants) | 12 | 6
  Week 14 (T4) | 0.71 (0.23) | 0.83 (0.46)

45. Other Pre Specified Outcome: Participant Satisfaction With VC-CBCS Telehealth Session Mean Score
Description: After intervention week 1 and week 14, participants in the VC-CBCS intervention completed a 15-item acceptability/satisfaction survey about their satisfaction with using telehealth sessions. Items were scored on a scale from 1= strongly disagree to 5=strongly agree. The average Total Telehealth Satisfaction score from week 1 and week 14 was created, which ranged from 1 to 5 with higher scores indicating greater satisfaction. A previously developed Telehealth Patient Satisfaction Questionnaire was modified for this study.
Time Frame: Baseline (T1) to Week 14 (T4)
Population: Participants randomized to Standard of Care received no intervention and did not complete survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VC-CBCS Intervention
Number analyzed (Participants) | 19
score on a scale
  Week 1 | 3.91 (0.68)
  Week 14 | 4.5 (0.38)

ADVERSE EVENTS:
Time Frame: From the time of first intervention session through the last intervention session, an approximate total of 14 weeks.
Arm/Group | VC-CBCS Intervention | Standard of Care (SC)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/8
Other Adverse Events (participants affected / at risk) | 0/21 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VC-CBCS Intervention (N=21) | Standard of Care (SC) (N=8)
Transient Ischemic Attack (TIA) (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04198584/Prot_SAP_000.pdf